CLINICAL TRIAL: NCT05444946
Title: A Randomized Controlled Trial to Compare Oral Itraconazole Versus Combination of Systemic Glucorticoids and Oral Itraconazole in Chronic Pulmonary and Allergic Bronchopulmonary Aspergillosis Overlap Syndrome
Brief Title: Oral Itraconazole Versus Combination of Systemic Glucorticoids and Oral Itraconazole in CPA-ABPA Overlap Syndrome
Acronym: GLITZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2021/SPL-749
Record Dates: First submitted 2022-06-21; First posted 2022-07-06 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pulmonary Aspergillosis; Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — Prednisone; Itraconazole

STUDY DESIGN:
Intervention Model Description: Subjects with CPA-ABPA overlap will be randomized to receive either a combination of systemic steroids and oral itraconazole or oral itraconazole alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid itraconazole (Experimental): Combination of oral glucocorticoid (prednisolone 0.5 mg/Kg body weight tapered over 4 months) and itraconazole for 12 months
  Interventions: Drug: Prednisone tablet and Itraconazole
- Itraconazole (Active Comparator): Oral itraconazole for 12 months
  Interventions: Drug: Oral itraconazole

INTERVENTIONS:
Drug: Prednisone tablet and Itraconazole — Oral prednisolone 0.5 mg/Kg body weight tapered over 4 months and oral itraconazole (400 mg/day). The dose of itraconazole will be adjusted according to therapeutic drug monitoring to achieve a serum trough level of 0.5 microgram/mL. traconazole will be given for 12 months
  Other Names: sporanox
  Arms: Steroid itraconazole
Drug: Oral itraconazole — Oral itraconazole (400 mg/day). The dose of itraconazole will be adjusted according to therapeutic drug monitoring to achieve a serum trough level of 0.5 microgram/mL. Itraconazole will be given for 12 months
  Other Names: sporanox
  Arms: Itraconazole

SUMMARY:
While ABPA and CPA represent two distinct manifestations of Aspergillus-related lung disease, there is an overlap of investigations that are currently used for the diagnosis of these entities. In a previous study, the authors have demonstrated that 22% of subjects with CPA fulfilled the obligatory criteria for ABPA. While the preferable therapy in patients with ABPA is systemic glucocorticoids, the primary therapy in CPA is oral triazoles. However, a different management protocol in the "overlap group" with low doses of glucocorticoids and triazoles, needs to be systematically explored. In this study the investigators intend to compare the clinical outcomes in subjects with ABPA-CPA overlap treated either with oral azoles or a combination of systemic glucocorticoids and oral azoles.

DETAILED DESCRIPTION:
Aspergillus causes a variety of pulmonary disorders depending on the host immunity. In immunocompetent hosts, it can cause allergic diseases, the prototype being allergic bronchopulmonary aspergillosis (ABPA). In immunosuppressed host, it causes life-threatening invasive disease. Chronic pulmonary aspergillosis (CPA) represents chronic Aspergillus infection of the pulmonary parenchyma in subjects with normal or slightly suppressed immunity, and generally an underlying structural lung disease (previously treated pulmonary tuberculosis, chronic obstructive pulmonary disease, sarcoidosis, diffuse parenchymal lung disease and others). The diagnosis of CPA is based on the presence of clinical symptoms (low-grade fever, weight loss, malaise, chronic cough, recurrent hemoptysis and others), radiological features (combination of one or more cavities and presence of fungal ball or fibrosis, pericavitary infiltrates, consolidation, nodules and pleural thickening) and the demonstration of either direct (growth of Aspergillus on sputum or bronchoalveolar lavage fluid [BALF] culture) or indirect (elevated serum or BALF galactomannan index or A.fumigatus-specific IgG or precipitin in serum) evidence of Aspergillus infection. Primarily seen in patients with asthma and cystic fibrosis, the diagnosis of ABPA is currently made on the combination of clinical (low grade fever, hemoptysis and others), radiological (bronchiectasis, mucus impaction, centrilobular nodules and others) and immunological (A.fumigatus-specific IgE and IgG, total IgE, and elevated eosinophils) findings.

While ABPA and CPA represent two distinct manifestations of Aspergillus-related lung disease, there is an overlap of investigations that are currently used for the diagnosis of these entities. For example, A.fumigatus-specific IgG and Aspergillus precipitins are used both in diagnosing ABPA and CPA.(10) The culture of respiratory tract secretions can demonstrate the growth of Aspergillus in both these disorders. Also, ABPA is a predisposing condition for developing CPA and it is likely that both ABPA and CPA may coexist. In a previous study, the authors have demonstrated that 22% of subjects with CPA fulfilled the obligatory criteria for ABPA. While CPA is primarily due to dysfunction of Th-1 immunity, ABPA represents an inflammatory response due to Th-2 hyper response. Thus, it is possible that subjects with ABPA-CPA overlap could have components of both heightened inflammatory response and local immune dysfunction thereby perpetuating structural lung damage. While the preferable therapy in patients with ABPA is systemic glucocorticoids, the primary therapy in CPA is oral triazoles. However, a different management protocol in the "overlap group" with low doses of glucocorticoids and triazoles, needs to be systematically explored. In this study the investigators intend to compare the clinical outcomes in subjects with ABPA-CPA overlap treated either with oral azoles or a combination of systemic glucocorticoids and oral azoles.

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfil criteria for ABPA and CPA as below.

The criteria for CPA would include the presence of all the following: (i) one or more clinical symptoms (persistent cough, recurrent hemoptysis, weight loss, malaise, fever and dyspnea) for ≥3 months; (ii) slowly progressive or persistent findings (one or more cavities and surrounding fibrosis, infiltrates, consolidation, with or without fungal ball or progressive pleural thickening) on computed tomography (CT) of the thorax; (iii) immunological (A.fumigatus-specific IgG >27 mgA/L or positive Aspergillus precipitins) or microbiological evidence of Aspergillus infection (growth of Aspergillus in respiratory secretions) and, (iv) exclusion of other pulmonary disorders with similar presentation.

The diagnosis of ABPA will be made based on the presence of all the following: (a) A.fumigatus specific IgE >0.35 kUA/L; (b) total IgE ≥500 IU/mL; (c) eosinophil count ≥500 cells/µL); (d) A.fumigatus IgG>27 mgA/L.

Exclusion Criteria:

(i) failure to provide informed consent; (ii) patients on immunosuppressive drugs, intake of prednisolone (or equivalent) >10 mg for at least 3 weeks or a diagnosis of human immunodeficiency virus syndrome; (iii) intake of antifungal triazoles for >3 weeks in the preceding three months; (iv) subjects with active pulmonary infection due to mycobacterium tuberculosis or mycobacteria other than tuberculosis (MOTT); (v) subjects with others forms of pulmonary aspergillosis (subacute and acute invasive aspergillosis); and, (vi) pregnancy.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Favourable response at six months after the randomization | 6 months after randomization
  Proportion of subjects with an overall favourable response at six months after the randomization. The overall response will be categorized as favourable: improved or stable clinical response with radiologically improved or stable disease

SECONDARY OUTCOMES:
Overall favourable response at 12 months after randomization | 12 months after randomization
  Proportion of subjects with an overall favourable response at 12 months after the randomization. The overall response will be categorized as favourable: improved or stable clinical response with radiologically improved or stable disease
frequency of relapses at 18-months after randomization | 18 months after randomization
  Relapse: will be defined as persistent worsening of symptoms (for 14 days or more) as measured by VAS and radiological worsening. The subjects will be investigated for other causes of worsening such as bacterial infection or reinfection/reactivation of tuberculosis before labelling the worsening due to relapse of CPA. A relapse will be defined as an event that occurs 3 months after stopping treatment
adverse events in either arm | 12 months after randomization
  Adverse events due to systemic glucocorticoids and oral itraconazole will be assessed at 2 weeks after treatment initiation and then at 3 months interval till treatment completion
Serum total IgE response to treatment | 6 weeks after treatment initiation
  proportion of subjects with 25% reduction in serum IgE at 6 weeks after treatment initiation
Serum total IgE during relapse | 18 months after randomization
  Proportion of subjects with 50% increase in serum IgE during relapse

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Chest clinic, PGIMER, Chandigarh
  - Chest clinic, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on email to the corresponding author